CLINICAL TRIAL: NCT00784186
Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Mid-trimester Termination of Pregnancy (14 - 21 Weeks LMP): A Randomized-controlled Double-blinded Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.3.1
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Abortion, Induced
Keywords: Pregnancy termination; abortion; medical abortion; 2nd trimester; mifepristone; misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mifepristone+misoprostol (Experimental): 200 mg mifepristone followed by 800 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses.
  Interventions: Drug: mifepristone+misoprostol; Drug: misoprostol
- misoprostol (Experimental): 800 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses.
  Interventions: Drug: misoprostol; Drug: placebo

INTERVENTIONS:
Drug: mifepristone+misoprostol — single dose of 200 mg mifepristone followed 24 hours later by 800 mcg misoprostol administered buccally and repeated every 3 hours for a maximum of 5 doses.
  Arms: mifepristone+misoprostol
Drug: misoprostol — placebo resembling mifepristone followed 24 hours later by 800 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses.
Drug: placebo — placebo resembling mifepristone taken 24 hours before 800 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses.
  Arms: misoprostol

SUMMARY:
The primary goal of this study is to determine the clinical advantage of pre-treatment with mifepristone in second trimester misoprostol induction abortion. This will be a randomized controlled double-blinded trial of 260 women comparing misoprostol alone to mifepristone plus misoprostol for second trimester (14-21 weeks' LMP) medical abortion.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 21 weeks gestation, based on menstrual history and clinical exam (with or without ultrasound)
* Meet legal criteria to obtain abortion
* Present with closed cervical os and no vaginal bleeding
* Live fetus at time of presentation for service
* Have no contraindications to study procedures, according to provider
* Be able to consent to procedure, either by reading consent document or by having consent document read to her
* Be willing to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Any contraindications to vaginal delivery, including placenta previa
* Presentation in active labor (defined as moderate to severe contractions every 10 minutes or less)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion: defined as complete evacuation using study drug without recourse to any additional intervention. | 24 hours

SECONDARY OUTCOMES:
Rate of fetal expulsion: defined as fetal expulsion with study drug alone. | 24 hours
Induction-to-abortion interval | Time elapsed between administration of the first misoprostol dose until expulsion of the fetus.
Total dose of misoprostol. | Assessed at time of complete abortion with study drug alone or when total maximum dose given.
Pain experienced by the woman as self-reported. | Assessed during exit interview.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, Principal Investigator — Gynuity Health Projects
Locations (2):
- Vietnam (2):
  - National Ob-Gyn Hospital, Hanoi
  - Hung Vuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Ngoc NTN, Shochet T, Raghavan S, Blum J, Nga NTB, Minh NTH, Phan VQ, Winikoff B. Mifepristone and misoprostol compared with misoprostol alone for second-trimester abortion: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):601-608. doi: 10.1097/AOG.0b013e318227214e. PMID 21860289